CLINICAL TRIAL: NCT06467760
Title: Thumb Hemi-Arthroplasty With Natural Kinematics; a Prospective Multicenter Study to Confirm the Safety and Efficacy of the InDx Implant
Acronym: THANKS PRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loci Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InDx03
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: CMC Joint Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device Implantation (Experimental): Single arm study - Device implanted
  Interventions: Device: InDx CMC Implant

INTERVENTIONS:
Device: InDx CMC Implant — The InDx CMC Implant is a hemiarthroplasty device for the CMC joint which consists of a unified assembly of three components: metacarpal stem, polyethylene liner, and articulating head. Because the device functions as a hemiarthroplasty, it does not link or constrain the CMC joint

SUMMARY:
Prospective, multicentric non-comparative confirmatory study to evaluate the safety and performance of the InDx CMC implant for the treatment of CMC joint arthritis.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age;
* The patient has a confirmed Grade I-III osteoarthritis of the CMC joint on clinical examination and X-ray;
* The patient is eligible for surgical treatment of CMC I arthrosis in the opinion of the investigator.
* The patient agrees to abstain from enrolment in any other clinical trials that will conflict or interfere with the interpretation of the results of this study, in the opinion of the Investigator, for the duration of the study;
* The patient is able to understand the aims and objectives of the trial and is willing to consent;
* The patient is willing and able to return for all study-related follow-up procedures;
* If the patient is female, is either using contraception or is postmenopausal, or male partner is using contraception

Exclusion Criteria:

* The patient is suffering from Rheumatoid arthritis in the index hand;
* The patient is suffering from Grade IV osteoarthritis of the CMC joint;
* The patient is suffering post-traumatic arthritis of the CMC joint in the index hand;
* The patient is a pregnant/lactating female (tested as per institutional requirements);
* Active or latent infection, or sepsis;
* Insufficient quantity or quality of bone and/or soft tissue in the index hand;
* Metal or polymer material sensitivity;
* Muscular imbalance, peripheral vascular disease that prohibits adequate healing, or a poor soft-tissue envelope in the surgical field, absence of musculoligamentous supporting structures, or peripheral neuropathy;
* Patient with previous thumb surgery in the index hand
* In the opinion of the investigator, any medical condition that makes the subject unsuitable for inclusion in the study, including, but not limited to

  * Patients with a diagnosis of concomitant injury that may interfere with healing
  * Patients with clinically significant renal, hepatic, cardiac, endocrine, hematologic, autoimmune, or any systemic disease or systemic infection that may make interpretation of the results difficult
* Patients who have undergone systemic administration within 30 days prior to implantation of any type of corticosteroid, antineoplastic, immunostimulating, or immunosuppressive agents
* Comorbidity that reduces life expectancy to less than 36 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Device Safety | 6 Months
  Determine the incidence of device failure, encompassing mechanical malfunction, structural compromise, loss of functionality due to device failure, or any deviation from the device's intended medical purpose. This will involve monitoring for adverse events requiring total revision surgery, or premature termination of device usage due to device failure.
Performance | 12 Months
  Measure the improvement in hand and wrist functionality using the Disabilities of the Arm, Shoulder, and Hand (DASH) score.
Performance | 12 Months
  Measure the improvement in hand and wrist functionality using the Patient-Rated Wrist/Hand Evaluation (PRWHE)

CONTACTS AND LOCATIONS:
Locations (1):
- Az Sint-Jan Brugge AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: Undecided